CLINICAL TRIAL: NCT06964217
Title: Overall Fracture Risk Immediately After Anti-hypertensive Medication Initiation and Temporal Trend in Initial Pharmacotherapy Regimens: An Observational Study
Brief Title: Immediate Fracture Risk After Antihypertensive Drug Initiation
Acronym: FADI
Status: Not yet recruiting | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Min Lee, Teaching Assistant (M.D), Ajou University School of Medicine
Other Study IDs: AJOUIRB-EX-2025-198
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Fracture
MeSH Terms: conditions — Hypertension; Fractures, Bone | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Monotherapy: Community-dwelling patients who get prescription of per oral anti-hypertensive drug (AHD) at an outpatient visit for hypertension diagnosis, without an exposure to any antihypertensive medication in the preceding year.
  Interventions: Drug: Monotherapy
- Combination therapy: Community-dwelling patients who get prescription of per oral antihypertensive pill/pills with two or more drug classes of AHDs - on a same day at an outpatient visit for hypertension diagnosis, without an exposure to any antihypertensive medication in the preceding year.
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: Monotherapy — Antihypertensive medications, regardless of dose or formulation, will be classified by their pharmacologic class. A total of eight drug classes will be considered: angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers (ARBs), beta-blockers, dihydropyridine calcium channel blockers (DHP-CCBs), non-dihydropyridine calcium channel blockers (non-DHP-CCBs), loop diuretics, thiazide and thiazide-like diuretics, and potassium-sparing diuretics.
  Exposure groups will be defined as follows:
  * Monotherapy: prescription of a single antihypertensive drug class on the index date.
  * Dual therapy: prescription of two ore more antihypertensive drug classes on the same index date.
  To qualify for group assignment, all drugs must be initiated on the same day, and the drug of interest is limited to the class described in group/cohort.
  Out of the two, this intervention will be monotherapy.
  Groups: Monotherapy
Drug: Combination therapy — Antihypertensive medications, regardless of dose or formulation, will be classified by their pharmacologic class. A total of eight drug classes will be considered: angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers (ARBs), beta-blockers, dihydropyridine calcium channel blockers (DHP-CCBs), non-dihydropyridine calcium channel blockers (non-DHP-CCBs), loop diuretics, thiazide and thiazide-like diuretics, and potassium-sparing diuretics.
  Exposure groups will be defined as follows:
  * Monotherapy: prescription of a single antihypertensive drug class on the index date.
  * Dual therapy: prescription of two or more antihypertensive drug classes on the same index date.
  To qualify for group assignment, all drugs must be initiated on the same day, and the drug of interest is limited to the class described in group/cohort.
  Out of the two, this intervention will be combination therapy.
  Groups: Combination therapy

SUMMARY:
This retrospective observational study aims to evaluate the short-term fracture risk associated with anti-hypertensive medication initiation using a self-controlled case series (SCCS) design and investigate temporal trends of initial anti-hypertensive regimen (monotherapy vs combination therapy) and subsequent fracture incidence. The investigators use the Korean Health Insurance Review and Assessment (HIRA) database to identify adults aged ≥65 with a new prescription for anti-hypertensive therapy and at least one incident non-traumatic fracture.

In the SCCS analysis, the investigators estimate the within-person incidence rate of overall fractures during the 30-day period following anti-hypertensive initiation compared to control periods. Temporal trends will be recorded through 2013 - 2022.

The primary outcome is overall non-traumatic fracture occurrence; the secondary outcome is incident proximal hip fracture. These outcomes are defined using diagnostic and procedural codes validated for use in claims data. This study aims to quantify both the immediate temporal association between treatment initiation and fracture risk, and the comparative safety of different initial anti-hypertensive regimens.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with at least 365 days of continuous observation prior to the index date (defined as the date of first antihypertensive medication prescription), with no prior antihypertensive use during that period
* At least one diagnosis of hypertension (ICD-10 codes I10-I13, I15) recorded within 180 days before the index date

Exclusion Criteria (main cohort):

* Any of the following occurring in the 365 days prior to the index date: Hospitalization (inpatient admission, including long-term care facility), transport-related trauma (ICD-10 codes V01-V99), Intentional self-harm (ICD-10 codes X60-X84, Y87), History of pathological fractures (e.g., M84.4, M90.7), Evidence of end-stage renal disease (ESRD), dialysis, kidney transplant, renal osteodystrophy

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling patients who are new users of antihypertensive medication, defined as individuals with no prior antihypertensive exposure in the 365 days prior to the index date
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall fracture risk | 45 days after initiation of antihypertensive medication
  First incidence of non-traumatic fracture in either proximal humerus, distal radius/ulna, thoraco-lumbar vertebrae, sacrum/pelvis, or proximal hip

SECONDARY OUTCOMES:
Hip fracture | 45 days after initiation of antihypertensive medication
  First incidence of non-traumatic proximal hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Rae Woong Park, M.D., Ph.D., Principal Investigator — Department of Biomedical Informatics, Ajou University School of Medicine, Suwon, Republic of Korea

IPD SHARING:
Plan to Share IPD: No
This study uses de-identified secondary data from the Korean Health Insurance Review and Assessment (HIRA) database. Individual-level data cannot be shared publicly due to legal and privacy restrictions.

REFERENCES:
- [Background] Butt DA, Mamdani M, Austin PC, Tu K, Gomes T, Glazier RH. The risk of hip fracture after initiating antihypertensive drugs in the elderly. Arch Intern Med. 2012 Dec 10;172(22):1739-44. doi: 10.1001/2013.jamainternmed.469. PMID 23165923
- [Background] Dave CV, Li Y, Steinman MA, Lee SJ, Liu X, Jing B, Graham LA, Marcum ZA, Fung KZ, Odden MC. Antihypertensive Medication and Fracture Risk in Older Veterans Health Administration Nursing Home Residents. JAMA Intern Med. 2024 Jun 1;184(6):661-669. doi: 10.1001/jamainternmed.2024.0507. PMID 38648065